CLINICAL TRIAL: NCT03004339
Title: A Phase 1 Randomized, Placebo and Active Comparator-controlled Trial, Double-blind for the IPs, Observer-blind for the Active Comparator, to Assess the Potency of SOR007 (Uncoated Nanoparticle Paclitaxel) Ointment in a Psoriasis Plaque Test
Brief Title: Trial to Assess the Potency of SOR007 Ointment in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DFB Soria, LLC (Industry)
Collaborators: Bioskin GmbH (Industry); US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOR007-2016-01
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SOR007 Ointment 2.0% (Experimental): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: SOR007 Ointment 2.0%
- SOR007 Ointment 1.0% (Experimental): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: SOR007 Ointment 1.0%
- SOR007 Ointment 0.3% (Experimental): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: SOR007 Ointment 0.3%
- SOR007 Ointment 0.15% (Experimental): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: SOR007 Ointment 0.15%
- SOR007 Ointment Placebo (Placebo Comparator): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: SOR007 Ointment Placebo
- Taclonex® Ointment (Active Comparator): Topical application once daily during a 12-day treatment period (10 treatments)
  Interventions: Drug: Taclonex® Ointment

INTERVENTIONS:
Drug: SOR007 Ointment 2.0%
  Arms: SOR007 Ointment 2.0%
Drug: SOR007 Ointment 1.0%
  Arms: SOR007 Ointment 1.0%
Drug: SOR007 Ointment 0.3%
  Arms: SOR007 Ointment 0.3%
Drug: SOR007 Ointment 0.15%
  Arms: SOR007 Ointment 0.15%
Drug: SOR007 Ointment Placebo
  Arms: SOR007 Ointment Placebo
Drug: Taclonex® Ointment
  Other Names: calcipotriene 0.005%/betamethasone dipropionate 0.064%
  Arms: Taclonex® Ointment

SUMMARY:
Evaluation of safety, pharmacokinetics, and anti-psoriatic efficacy to assess SOR007 Ointment in topical formulations

DETAILED DESCRIPTION:
This is a two-center, randomized, placebo- and active comparator-controlled trial that will be double-blind for the investigational products (IPs) and observer-blind for the active comparator with intra-individual comparison of treatments. Twelve male and post-menopausal female volunteer subjects, aged 18 years or older, with psoriasis vulgaris and mild or moderate chronic plaque(s) in a stable phase and an area sufficient for six treatment fields, will be enrolled. SOR007 Ointment will be administered topically at four concentrations (0.15%, 0.3%, 1%, and 2%), in addition to a placebo ointment (SOR007 without the active pharmaceutical ingredient) and an active comparator, Taclonex® Ointment (calcipotriene 0.005 % and betamethasone dipropionate 0.064 %). Treatments will be administered once daily, 10 times over a 12-day trial period. Assessments will include safety, pharmacokinetics (PK), and preliminary efficacy as determined by measurement of psoriatic infiltrate using 22-megahertz (MHz) sonography as well as clinical scoring on a 5-point scale. Subjects who withdraw early for reasons unrelated to investigational product adverse events (AEs) will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* men and surgically sterile or post-menopausal (at least since 12 months amenorrhoea) women aged 18 years or older. The non-childbearing potential of women needs to be confirmed by medical record or in writing by a gynecologist, if that is not possible a follicle stimulating hormone (FSH) test will be performed on female subjects to confirm menopause, unless they are receiving hormonal replacement therapy for treatment of menopause symptoms;
* subjects with psoriasis vulgaris in a chronic stable phase and mild to moderate plaque(s) with up to three plaque areas sufficient for six treatment fields;
* the target lesion(s) should be on the trunk or extremities (excluding palms/soles); psoriatic lesion on the knees or elbows are not to be used as a target lesion;
* plaques to be treated should have a comparable psoriatic infiltrate thickness of at least 200 μm;
* the physical examination of the skin must be without disease findings other than psoriasis vulgaris unless the investigator considers an abnormality to be irrelevant to the outcome of the clinical trial;
* male volunteers must agree to sexual abstinence or use adequate contraception when sexually active in combination with their female partners, if they are of childbearing potential. That means the volunteer must be vasectomized or use a condom and his female partner must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 % per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, or non-DalKon Shield intra-uterine devices [IUDs]. This applies from signing of the informed consent form until 90 days after the last study drug administration. Methods of contraception must have been effective for at least 30 days on the day of signing the informed consent form. Male volunteers must also refrain from sperm donation from signing of the informed consent form until 90 days after the last study drug administration;
* written informed consent obtained.

Exclusion Criteria:

* pregnancy and nursing;
* other skin disease or condition noted on physical examination that is considered by the investigator to be relevant to the outcome of the trial;
* subjects with acute psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica and pustular psoriasis;
* any topical antipsoriatics on plaques potentially to be treated in this trial (including corticosteroids, vitamin D analogues, immunomodulators, retinoids, dithranol and tar, except for salicylic acid and except for treatment on the face, ears and scalp) in the 4 weeks before first treatment and/or during the trial;
* systemic treatment with antipsoriatics e.g. corticosteroids, cytostatics, retinoids, dimethylfumarate in the three months before first treatment and during the trial;
* systemic treatment with biological treatments: ustekinumab or secukinumab within six months or adalimumab, infliximab and etanercept within three months before first treatment and during the trial;
* UV-therapy within four weeks before first treatment and during the trial;
* treatment with systemic or locally acting medications which might have countered or influenced the trial aim (medications which are known to provoke or aggravate psoriasis, e.g. antimalarial drugs, lithium) within eight weeks before first treatment and/or during the trial. Beta-blockers or angiotensin-converting enzyme (ACE) inhibitors are allowed if on a stable dose for 3 months before study medication initiation;
* intake of Anticoagulant Drugs, e.g. Warfarin, Coumadin. Antiplatelet Drugs e.g. Acetyl salicylic acid are permitted unless considered contraindicated by the investigator for blood withdrawal for PK analyses;
* known allergic reactions, irritations or sensitivity to the active ingredients or other components of the IPs;
* known allergic reactions, irritations or sensitivity to the comparator's active ingredient and/or components;
* contraindications according to summary of product characteristics of the active comparator;
* evidence of drug or alcohol abuse;
* symptoms of a clinically significant illness that may place the subject at risk by trial participation or influence the outcome of the trial in the four weeks before first treatment and during the trial;
* participation in the treatment phase of another clinical trial within the last four weeks prior to first treatment in this clinical trial;
* in the opinion of the investigator or physician performing the initial examination the subject should not participate in the trial, e.g. due to probable noncompliance or inability to understand the trial and give adequately informed consent;
* close affiliation with the investigator (e.g. a close relative) or persons working at bioskin GmbH or Modoc or subject is an employee of sponsor;
* subject is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Change in the thickness of the echolucent band (ELB) | 12 days

SECONDARY OUTCOMES:
Evaluation of the antipsoriatic efficacy by clinical assessment using a 5-point score | 12 days

OTHER OUTCOMES:
Safety analysis: Summary of Treatment-Emergent Adverse Events | 26 days
  Treatment-emergent adverse events (TEAEs), i.e. AEs with an onset or worsening on or after the time of the first investigational product (IP) application, will be reported. TEAEs will be summarized by the number of subjects reporting TEAEs, primary system organ class (SOC), preferred term (PT), severity, and relationship to IP. Summaries will be provided by the relation to a specific treatment test field or as not related to a specific test field. Vital signs parameters will be summarized descriptively by treatment and visit, including changes from screening visit. Only clinical relevance will be listed.
Pharmacokinetic analysis: Maximum Plasma Concentration of Paclitaxel (Cmax) | 12 days
  PK levels of paclitaxel in the plasma will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Gere S diZerega, MD, Study Chair — US Biotest, Inc./DFB Soria, LLC
Locations (2):
- United States (2):
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., College Station, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parisi R, Symmons DP, Griffiths CE, Ashcroft DM; Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013 Feb;133(2):377-85. doi: 10.1038/jid.2012.339. Epub 2012 Sep 27. PMID 23014338
- [Background] Nestle FO, Di Meglio P, Qin JZ, Nickoloff BJ. Skin immune sentinels in health and disease. Nat Rev Immunol. 2009 Oct;9(10):679-91. doi: 10.1038/nri2622. Epub 2009 Sep 18. PMID 19763149
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Schiff PB, Horwitz SB. Taxol stabilizes microtubules in mouse fibroblast cells. Proc Natl Acad Sci U S A. 1980 Mar;77(3):1561-5. doi: 10.1073/pnas.77.3.1561. PMID 6103535
- [Background] Mirzapoiazova T, Kolosova IA, Moreno L, Sammani S, Garcia JG, Verin AD. Suppression of endotoxin-induced inflammation by taxol. Eur Respir J. 2007 Sep;30(3):429-35. doi: 10.1183/09031936.00154206. Epub 2007 May 30. PMID 17537765
- [Background] Zhang L, Dermawan K, Jin M, Liu R, Zheng H, Xu L, Zhang Y, Cai Y, Chu Y, Xiong S. Differential impairment of regulatory T cells rather than effector T cells by paclitaxel-based chemotherapy. Clin Immunol. 2008 Nov;129(2):219-29. doi: 10.1016/j.clim.2008.07.013. Epub 2008 Sep 3. PMID 18771959
- [Background] Belotti D, Vergani V, Drudis T, Borsotti P, Pitelli MR, Viale G, Giavazzi R, Taraboletti G. The microtubule-affecting drug paclitaxel has antiangiogenic activity. Clin Cancer Res. 1996 Nov;2(11):1843-9. PMID 9816139
- [Background] Ehrlich A, Booher S, Becerra Y, Borris DL, Figg WD, Turner ML, Blauvelt A. Micellar paclitaxel improves severe psoriasis in a prospective phase II pilot study. J Am Acad Dermatol. 2004 Apr;50(4):533-40. doi: 10.1016/j.jaad.2003.09.018. PMID 15034502
- [Background] Dumas KJ, Scholtz JR. The psoriasis bio-assay for topical corticosteroid activity. Acta Derm Venereol. 1972;52(1):43-8. No abstract available. PMID 4111105
- [Background] Bangha E, Elsner P. Evaluation of topical antipsoriatic treatment by chromametry, visiometry and 20-MHz ultrasound in the psoriasis plaque test. Skin Pharmacol. 1996;9(5):298-306. doi: 10.1159/000211428. PMID 8990504
- [Background] Kvist PH, Svensson L, Hagberg O, Hoffmann V, Kemp K, Ropke MA. Comparison of the effects of vitamin D products in a psoriasis plaque test and a murine psoriasis xenograft model. J Transl Med. 2009 Dec 17;7:107. doi: 10.1186/1479-5876-7-107. PMID 20017943
- [Background] Kragballe K, Noerrelund KL, Lui H, Ortonne JP, Wozel G, Uurasmaa T, Fleming C, Estebaranz JL, Hanssen LI, Persson LM. Efficacy of once-daily treatment regimens with calcipotriol/betamethasone dipropionate ointment and calcipotriol ointment in psoriasis vulgaris. Br J Dermatol. 2004 Jun;150(6):1167-73. doi: 10.1111/j.1365-2133.2004.05986.x. PMID 15214905
- [Background] Kaufmann R, Bibby AJ, Bissonnette R, Cambazard F, Chu AC, Decroix J, Douglas WS, Lowson D, Mascaro JM, Murphy GM, Stymne B. A new calcipotriol/betamethasone dipropionate formulation (Daivobet) is an effective once-daily treatment for psoriasis vulgaris. Dermatology. 2002;205(4):389-93. doi: 10.1159/000066440. PMID 12444337
- [Background] Reich K, Bewley A. What is new in topical therapy for psoriasis? J Eur Acad Dermatol Venereol. 2011 Jun;25 Suppl 4:15-20. doi: 10.1111/j.1468-3083.2011.04061.x. PMID 21507079
- [Background] Schmid-Ott G, Kunsebeck HW, Jager B, Sittig U, Hofste N, Ott R, Malewski P, Lamprecht F. Significance of the stigmatization experience of psoriasis patients: a 1-year follow-up of the illness and its psychosocial consequences in men and women. Acta Derm Venereol. 2005;85(1):27-32. doi: 10.1080/000155550410021583. PMID 15848987
- [Background] Gupta MA, Gupta AK. Age and gender differences in the impact of psoriasis on quality of life. Int J Dermatol. 1995 Oct;34(10):700-3. doi: 10.1111/j.1365-4362.1995.tb04656.x. PMID 8537157
- [Background] Remitz A, Reitamo S, Erkko P, Granlund H, Lauerma AI. Tacrolimus ointment improves psoriasis in a microplaque assay. Br J Dermatol. 1999 Jul;141(1):103-7. doi: 10.1046/j.1365-2133.1999.02927.x. PMID 10417522